CLINICAL TRIAL: NCT03204357
Title: Targeted Fresh Autologous Whole Blood Transfusion After Cardiopulmonary Bypass: a Prospective Randomized Controlled Trial.
Brief Title: Fresh Autologous Whole Blood Transfusion After Cardiopulmonary Bypass
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-2647
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Disease; Bleeding Postoperative
Keywords: Cardiac surgery
MeSH Terms: conditions — Heart Diseases; Postoperative Hemorrhage

STUDY DESIGN:
Intervention Model Description: The study design is a prospective randomized interventional trial of transfusion of fresh autologous whole blood versus standard of care expectant management of bleeding during elective cardiac surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh Autologous whole blood transfusion (Experimental): The experimental group will have 15% of the estimated blood volume of autologous blood collected. This transfusion will be given at the end of the procedure.
  Interventions: Other: Fresh Autologous whole Blood
- Standard of Care Expectant Management of bleeding (Active Comparator): the control group that will receive the standard of care expectant management of bleeding and transfusion of allogenic banked blood products
  Interventions: Other: Standard of Care Expectant management of bleeding

INTERVENTIONS:
Other: Fresh Autologous whole Blood — Subjects randomized this arm will receive fresh autologous whole blood
  Arms: Fresh Autologous whole blood transfusion
Other: Standard of Care Expectant management of bleeding — the control group that will receive the standard of care expectant management of bleeding and transfusion of allogenic banked blood products
  Arms: Standard of Care Expectant Management of bleeding

SUMMARY:
Autologous blood transfused at the end of cardiopulmonary bypass will reduce total blood loss 24 hours after surgery and improve mitochondrial oxygen delivery measured by plasma succinate levels.

The study design is a prospective randomized interventional trial of transfusion of fresh autologous whole blood versus standard of care expectant management of bleeding during elective cardiac surgery.

DETAILED DESCRIPTION:
Cardiac surgery carries a significant risk of bleeding requiring transfusion of stored blood products and blood transfusion associated with cardiac surgery consumes 20% of the blood supply worldwide. Although transfusion may be life-saving, significant risks of complications such as lung injury or even an increase in mortality are associated with transfusion. Decreasing transfusion requirements during cardiac surgery has the potential to reduce the rate of complications, improve patient outcomes, and reduce cost resulting in increased value for both the patient and the health system as a whole. Collection of autologous blood before cardiopulmonary bypass (CPB) for transfusion after CPB has been shown to be both safe and effective for reducing blood loss during cardiac surgery, but this intervention has not been targeted to a patient population at high risk for bleeding and transfusion. Fresh whole blood has the capacity to restore coagulation system function during profound coagulopathy in a trauma setting or following massive transfusion by an unknown mechanism. One unit of fresh whole blood is able to restore clotting function equivalent to that achieved by 10 units of pooled platelets. Autologous whole blood collection prior to CPB for transfusion post-operatively has been shown to improve coagulation and decrease clot lysis but is not routinely performed because 90% to 95% of patients do not have extensive blood loss and subsequent coagulopathy. Coupling accurate pre-operative bleeding risk prediction with autologous fresh whole blood collection for transfusion after CPB would target an established, low cost, low risk intervention to an at risk patient population who may experience significant benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged 18 to 90
2. Able to provide informed consent
3. Willing to accept autologous or allogenic blood transfusion
4. Scheduled for elective cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

1. Pre-operative administration of allogenic blood bank products in the previous 3 months
2. Hemodynamically unstable defined as a systolic blood pressure less than 90 mmHg with a heart rate greater 100 or requiring intravenous vasopressor medications
3. Significant active infection or sepsis defined by positive blood culture or positive wound culture
4. Hemoglobin less than 7 g/dl

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Estimated Blood Loss | Within 24 hours after surgery
  Blood loss is estimated as a percent of total estimated blood volume in the first 24 hours after cardiac surgery.

SECONDARY OUTCOMES:
Number of allogenic transfusions given | 31 days
  Allogenic blood product transfusion requirements
Severity of peri-operative stroke | 31 days
  The severity of peri-operative stroke will be measured by the National institute of health stroke scale
Incident of peri-operative stroke | 31 days
  The incident of peri-operative stroke will be measured by the National institute of health stroke scale
Development of Post-operative delirium | 31 days
  Measured by Confusion Assessment Method - Intensive Care Unit
Development of Myocardial Infarction | 31 days
  As measured by physiological parameters
Development of Heart failure | 31 days
  As measured by physiological parameters
Detection of New Onset Atrial fibrillation | 31 days
  As measured by an electrocardiogram
Development of Lung injury | 31 days
  Measured by a Pa02/Fi02 ratio
Time to extubation | 31 days
  Time from when the breathing tube was placed to the time when the breathing tube is removed
Development of Acute Kidney Injury | 31 days
  As measured by abnormal lab values
Initiation of renal replacement therapy | 31 days
  Time to start of renal replacement therapy
ICU length of stay | 31 days
  This will be measured by the number of days in ICU
Evaluation of Vasopressor requirements (1) | 31 days
  Measurement of the amount of vasopressors given
Evaluation of Vasopressor requirements (2) | 31 days
  Measurement of the types of vasopressors given
Change in endothelial function measured by flow mediated dilation of the brachial artery | 24 hours after surgery
  Measurement of brachial artery dilation in response to flow by ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Clendenen, M.D., Principal Investigator — University of Colorado - School of Medicine
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No